CLINICAL TRIAL: NCT03243344
Title: Randomized Medico-economic Assessment of Preventive Devices Used for Post-operative Hemorrhagic Risk in Endonasal Surgery
Brief Title: Randomized Assessment of Devices Used to Prevent Post-operative Hemorrhagic Risk in Endonasal Surgery
Acronym: PRHEPOCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SHC/2009/001/P
Record Dates: First submitted 2017-08-02; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2010-03

CONDITIONS: Otorhinolaryngologic Diseases
MeSH Terms: conditions — Otorhinolaryngologic Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Surgiflo (Experimental): Using Surgiflo® (Absorbable Gelatin Hemostatic) for the post-operative haemostasis in endonasal surgery.
  Interventions: Device: Surgiflo
- Floseal (Experimental): Using Floseal® (Absorbable Gelatin Hemostatic) containing human thrombin for the post-operative haemostasis in endonasal surgery
  Interventions: Device: Floseal
- Algosteril (Experimental): Using Algosteril® (Hemostatic Sterile Wick) for the post-operative haemostasis in endonasal surgery
  Interventions: Device: Algosteril
- Abstention (No Intervention): Not using device for the post-operative haemostasis in endonasal surgery

INTERVENTIONS:
Device: Surgiflo — using device during the endonasal surgery.
  Arms: Surgiflo
Device: Floseal — using device during the endonasal surgery.
  Arms: Floseal
Device: Algosteril — using device during the endonasal surgery.
  Arms: Algosteril

SUMMARY:
This study evaluates the efficiency and the cost of three medical devices and the abstention of the use of specific product for the post-operative haemostasis in endonasal surgery .

DETAILED DESCRIPTION:
Surgiflo® is a matrix of haemostatic frost of porcine protein origin is the coverage of the post-operative bleeding of which one of the indications is in endonasal surgery.

Floseal® is a haemostatic frost(gel) containing of the thrombin.

Algosteril® is a lint tent of arginate of calcium.

ELIGIBILITY:
Inclusion Criteria:

* endonasal surgery schedule
* Surgical indications:

hypertrophic rhinitis, repeated or chronic infections, extraction of foreign body, polyposes naso-sinusal, benign tumors limited to the nasal pit and in sine,

Exclusion Criteria:

* Pregnant Woman
* Disorder of the haemostasis known or disrupted preoperative biological balance assessment
* Use of treatment disrupting the blood coagulation (anti platelet, anti vitamin K, AINS)
* Unchecked HTA by the treatment and/or preoperative > mmHg 160/90
* Surgical Act including a septoplasty
* malignant tumoral surgical Indication, or mild overtaking the naso-sinusial system
* Dacryocystorhinostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Per-operative hemostasis | Hours 0
  Time needs to observe hemostasis after the device set up
Hemostasis in the 6 first hours | Hours 6
  Number of compresses used from Hours 0 to Hours 6.
Hemostasis at the 24th hour | Hours 24
  * Algosteril arm (after having removed the wick): spontaneous observation of hemostasis in less that 3 min (yes/no) and needs to have a new intervention to stop bleedings (type)
  * Surgiflo, Floseal, Abstention arms: time to observe hemostasis if bleedings occurred.
Spontaneous hemorrhagic events | from Hours 0 to Day 45
  number of spontaneous hemorrhagic events.

SECONDARY OUTCOMES:
Preoperative assessment | Before the endonasal surgery
  Preoperative scanner assessment with Lund ans Mackay score
Preoperative assessment | Hours 0
  Laboratory tests of hemostasis (platelets, fibrinogen...)
Device evaluation by the surgeon | Hours 0
  time needs to set up the device
Device evaluation by the surgeon | Hours 0
  subjective assessment of the implementation ease

CONTACTS AND LOCATIONS:
Overall Officials: Laurent TAVERNIER, PH, Principal Investigator — CHU Besançon